CLINICAL TRIAL: NCT02155192
Title: Exploratory Genetic Study in Subjects With Moderate to Severe Psoriasis
Brief Title: An Exploratory Genetic Study in Participants With Psoriasis
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR103877; NOCOMPOUNDPSO0001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2014-06-02; First posted 2014-06-04 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Psoriasis
Keywords: CNTO1959PSO2001; C0743T08; C0743T09; C0743T12; Psoriasis; Pharmacogenomics
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Two buccal swab samples will be collected to extract Deoxyribonucleic acid (DNA).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Cohort 1: Participants who participated in NCT01483599 (X-PLORE) study.
  Interventions: Drug: No Intervention
- Cohort 2: Participants who participated in NCT00267969 (PHOENIX 1) study.
  Interventions: Drug: No Intervention
- Cohort 3: Participants who participated in NCT00307437 (PHOENIX-2) study.
  Interventions: Drug: No Intervention
- Cohort 4: Participants who participated in NCT00454584 (ACCEPT) study.
  Interventions: Drug: No Intervention

INTERVENTIONS:
Drug: No Intervention

SUMMARY:
The purpose of this study is to evaluate the association between genetic factors and response to treatment (guselkumab, ustekinumab, adalimumab, or etanercept) and psoriasis (scaly skin rash).

DETAILED DESCRIPTION:
This is a Phase 0, exploratory (intended to be conducted early in Phase 1, involve limited human exposure, have no therapeutic intent and are not intended to examine clinical tolerability), multicenter (when more than one hospital or medical school team work on a medical research study) and pharmacogenomics study in participants with psoriasis. Participants who were treated in study Phase 2 NCT01483599 (X-PLORE), Phase 3 NCT00267969 (PHOENIX 1), Phase 3 NCT00307437 (PHOENIX 2) or Phase 3 NCT00454584 (ACCEPT), will be returning to their study site where a deoxyribonucleic acid (DNA) sample will be obtained for pharmacogenomics assessment. There will be no follow-up beyond the study site visit.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have been randomly assigned and treated in the NCT01483599 (X-PLORE), NCT00267969 (PHOENIX 1), NCT00307437 (PHOENIX-2) , or NCT00454584 (ACCEPT) studies
* Sign an informed consent document indicating that they understand the purpose of and procedures required for this study and are willing to participate in this study

Exclusion Criteria:

* Participants has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the subject (for example, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who were treated in the CNTO1959PSO2001 study, C0743T08 study, C0743T09 or C0743T12 study will be assessed.
Sampling Method: Non-Probability Sample
Enrollment: 712 (Actual)
Dates: Start 2014-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Percentage of Responders With Association Between Clinical Response and Genetic Factor | Day 1
  Participants with clinical response from previous studies will be evaluated for the association with genetic factors (for example, human leukocyte antigen [HLA], Cw6 allele). Clinical response in previous studies were evaluated by psoriasis area and severity index (PASI) score: a widely used tool for the measurement of severity of psoriasis. This is a test of how bad a participant's psoriasis is. The scale combines redness, scaling, and thickness, as well as overall body involvement to determine the PASI score, scale ranges from 0 (best) to 72 (worst); and physician global assessment (PGA): The PGA is 6-point scale used in clinical trials of various diseases. In this the physician checks the state of the disease and gives them score from 0 (clear) to 5 (severe). Percentage of participants will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trials, Study Director — Janssen Research & Development, LLC
Locations (19):
- United States (12):
  - Bakersfield, California
  - Los Angeles, California
  - Ocala, Florida
  - Alpharetta, Georgia
  - Arlington Heights, Illinois
  - Indianapolis, Indiana
  - Louisville, Kentucky
  - Andover, Massachusetts
  - St Louis, Missouri
  - New York, New York
  - Portland, Oregon
  - Webster, Texas
- Canada (7):
  - Moncton, New Brunswick
  - Hamilton, Ontario
  - London, Ontario
  - Toronto, Ontario
  - Waterloo, Ontario
  - Montreal, Quebec
  - Québec, Quebec